CLINICAL TRIAL: NCT02454933
Title: A Phase III, Multi-Centre, Open Label, Randomized Study to Assess the Efficacy and Safety of AZD9291 in Combination With MEDI4736 Versus AZD9291 Monotherapy in Patients With Locally Advanced or Metastatic Epidermal Growth Factor Receptor T790M Mutation-positive Non-Small Cell Lung Cancer Who Have Received Prior Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy (CAURAL)
Brief Title: Study of AZD9291 Plus MEDI4736 Versus AZD9291 Monotherapy in NSCLC After Previous EGFR TKI Therapy in T790M Mutation Positive Tumours
Acronym: CAURAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5165C00001; 2015-001858-15 (EudraCT Number)
Record Dates: First submitted 2015-05-14; First posted 2015-05-27 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced or Metastatic EGFR T790M+ NSCLC
Keywords: Phase III Open Label Study; AZD9291 plus MEDI4736 versus AZD9291 Monotherapy; NSCLC After Previous EGFR TKI Therapy; T790M Mutation Positive Tumours.
MeSH Terms: interventions — osimertinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI4736 & AZD9291 Combination (Experimental): 10mg/kg q2w (IV) infusion & once daily tablet 80 mg
  Interventions: Drug: AZD9291; Drug: MEDI4736
- AZD9291 Monotherapy (Experimental): Once daily tablet 80 mg
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — Once daily tablet 80 mg
Drug: MEDI4736 — 10mg/kg q2w (IV) infusion
  Arms: MEDI4736 & AZD9291 Combination

SUMMARY:
A Phase III, Multi-Centre, Open Label, Randomized Study to Assess the Efficacy and Safety of AZD9291 in Combination with MEDI4736 versus AZD9291 Monotherapy in patients with Locally Advanced or Metastatic Epidermal Growth Factor Receptor T790M mutation-positive Non-Small Cell Lung Cancer who have received Prior Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy

DETAILED DESCRIPTION:
This a phase III, Multi Centre, Open Label, Randomized, Study to Assess the Efficacy and Safety of AZD9291 (80 mg, orally, once daily) in Combination with MEDI4736 (10 mg/kg (IV) infusion q2w) versus AZD9291 Monotherapy (80 mg, orally, once daily) in patients with a confirmed diagnosis of Epidermal Growth Factor Receptor (EGFR) T790M mutation positive NSCLC, who have progressed following prior therapy with an approved Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) agent. The randomization will be stratified by previous lines of treatment (2nd or 3rd+) and ethnicity (Asian or Non-Asian). A mandatory biopsy will be needed for central testing of T790M mutation status following confirmed disease progression on the most recent treatment regimen. The primary objective of the study is To investigate the safety and tolerability profile of AZD9291 in combination with MEDI4736.

350 patients were originally planned to be evaluated across the two below populations. The recruitment was stopped due to new information on safety of the combination, received from another trial in similar patient population

1. 2nd line: patients who have progressed following an approved first-line EGFR-TKI treatment but who have not received further treatment.
2. 3rd line or higher: patients who have progressed following prior therapy with an approved EGFR-TKI and an additional anti-cancer treatment. Patients may have also received additional lines of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years. Japan patients aged at least 20 years.
* Locally advanced/metastatic NSCLC, not amenable to curative surgery or radiotherapy
* Confirmation from a previous archival sample that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity
* Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI. Additional other lines of therapy may have been given. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.
* Patients must have central lab confirmation of tumour T790M status from a biopsy taken after disease progression on the most recent treatment regimen. Only patients with T790M+ will be included in the study
* At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥ 15mm) with computerised tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements
* World Health Organisation (WHO) performance status 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks
* Females of child-bearing potential using contraception; negative pregnancy test

Exclusion Criteria:

* Treatment with an EGFR-TKI within 5x half-life of study entry; any cytotoxic chemotherapy, investigational agents or other anticancer drugs within 14 days of study entry; current treatment with potent inhibitors/inducers of cytochrome P450 3A4 (CYP3A4); previous treatment with AZD9291 (or other agents specifically targeted against EGFR T790M mutation positive NSCLC); Prior neo-adjuvant or adjuvant chemotherapy treatment within 6 months of starting 1st EGFR TKI treatment; prior exposure to immune-mediated therapy including, but not limited to, other anti cytotoxic T-lymphocyte-associated antigen 4 (anti CTLA-4), anti- programmed cell death 1 (anti-PD-1), anti- programmed cell death ligand 1 (anti-PD-L1), and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines; radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks; major surgery within 4 weeks;
* Current or prior use of immunosuppressive medication within 14 days before the first dose of MEDI4736 (excluding intranasal, inhaled, topical steroids, or local steroid injections)
* Unresolved toxicities from prior therapy
* History of active primary immunodeficiency
* Unstable brain metastases or spinal cord compression
* Severe/uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant, bleeding diatheses or infection
* Cardiac disease
* Ophthalmological conditions
* Refractory nausea/vomiting, chronic gastrointestinal diseases or bowel resection
* Past history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* History of another primary malignancy
* Active or prior documented autoimmune or inflammatory disorders within the past 3 years prior to the start of treatment
* History of organ transplant that requires use of immunosuppressive medications
* Known history of tuberculosis
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of MEDI4736
* Inadequate bone marrow reserve or organ function

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horn, MD, Principal Investigator — Vanderbilt University, Nashville, USA; James CH Yang, MD, Principal Investigator — National Taiwan University Hospital
Locations (11):
- Research Site, Toronto, Ontario, Canada
- South Korea (7):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Ulsan
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: d5165c00001_CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3824&filename=d5165c00001_CSP.pdf
- See also: d5165c00001_SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3824&filename=d5165c00001_SAP.pdf
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5165C00001&attachmentIdentifier=6ca2ff84-5370-43f5-947d-78cc8acda613&fileName=d5165c00001-study-synopsis_CAURAL_CSR_synopsis_Redacted_with_correction.pdf&versionIdentifier=
- See also: CSR synopsis addendum — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5165C00001&attachmentIdentifier=6e0ef65b-c5cd-4551-a00b-f41d0e1a0f73&fileName=d5165c00001-Study_Report-Addendum_Synopsis_Jul2018_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited to this study in 9 centres in South Korea, Canada and Taiwan. First subject first visit: 26 August 2015.
Pre-assignment Details: 60 subjects with a confirmed diagnosis of Epidermal Growth Factor Receptor (EGFR) T790M mutation postive non-small cell lung cancer (Stage IIIB-IV) with progression following prior therapy with an approved EGFR tyrosine kinase inhibitor agent were screened, and 29 were assigned to treatment.
Groups:
- Osimertinib 80 mg: Subjects were randomised to receive osimertinib (AZD9291) monotherapy (80 milligrams [mg], orally, once daily).
- Osimertinib 80 mg + Durvalumab 10 mg/kg: Subjects were randomised to receive osimertinib 80 mg, orally, once daily in combination with durvalumab (MEDI4736) 10 mg/kilogram (mg/kg) intravenous (IV) infusion every 2 weeks.
Period: Overall Study
Arm/Group | Osimertinib 80 mg | Osimertinib 80 mg + Durvalumab 10 mg/kg
Started (Actual treatment received) | 17 | 12 (2 subjects switched to osimertinib monotherapy Cycle 1 Day 1)
Treatment Group Randomised to | 15 | 14
Ongoing at Primary Analysis Data Cut-off | 9 | 4
Completed (Subjects completing study at final analysis data cut-off) | 5 | 1
Not Completed | 12 | 11
Not completed — Progressive disease | 10 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all subjects who received at least one dose of randomised treatment.
Groups:
- Osimertinib 80 mg: Subjects were randomised to receive osimertinib (AZD9291) monotherapy (80 mg, orally, once daily).
- Osimertinib 80 mg + Durvalumab 10mg/kg: Subjects were randomised to receive osimertinib 80 mg, orally, once daily in combination with durvalumab (MEDI4736) 10 mg/kg IV infusion every 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Osimertinib 80 mg | Osimertinib 80 mg + Durvalumab 10mg/kg | Total
Number analyzed (Participants) | 17 | 12 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.6) | 57.6 (11.2) | 60.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 12 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 11 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs) as a Measure of the Safety and Tolerability of Osimertinib in Combination With Durvalumab
Description: As a measure of the safety and tolerability of osimertinib in combination with durvalumab the number of subjects who experienced any treatment emergent AE (TEAE), any causally related AE, any serious AE (SAE), and any causally related SAE are presented.
Time Frame: From Baseline up to primary analysis data cut-off (up to 24 months).
Population: The safety analysis set consisted of all subjects who received at least one dose of randomised treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib 80 mg + Durvalumab 10mg/kg
Number analyzed (Participants) | 12
Participants
  Any AE | 12
  Any AE causally related to treatment | 8
  Any AE causally related to osimertinib only | 8
  Any AE causally related to durvalumab only | 4
  Any AE causally related to osimertinib+durvalumab | 3
  Any SAE | 3
  Any SAE causally related to treatment | 1

ADVERSE EVENTS:
Time Frame: TEAEs are presented from the date of first dose and up to and including 30 days following the date of the last dose of osimertinib or 90 days following the date of last dose of durvalumab (up to approximately 31 months).
Description: The safety analysis set consisted of all subjects who received at least one dose of randomised treatment.
Groups:
- Osimertinib 80 mg + Durvalumab 10 mg/kg: Subjects were randomised to receive osimertinib 80 mg, orally, once daily in combination with durvalumab (MEDI4736) 10 mg/kg IV infusion every 2 weeks.
Arm/Group | Osimertinib 80 mg | Osimertinib 80 mg + Durvalumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 4/17 | 8/12
Serious Adverse Events (participants affected / at risk) | 6/17 | 3/12
Other Adverse Events (participants affected / at risk) | 17/17 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib 80 mg (N=17) | Osimertinib 80 mg + Durvalumab 10 mg/kg (N=12)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osimertinib 80 mg (N=17) | Osimertinib 80 mg + Durvalumab 10 mg/kg (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (35) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 2 (2)
Eyelid pain (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1)
Retinal drusen (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 8 (12) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 2 (4)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site injury (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2)
Complication associated with device (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (3) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 7 (10) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (4)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Vestibulitis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 4 (6) | 1 (2)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (5) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 2 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (6) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Renal vein embolism (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Uterine mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Xanthelasma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Subject enrolment was terminated early on 29 September 2015 after higher than anticipated incidence of interstitial lung disease-like events in subjects receiving osimertinib + durvalumab in a separate Phase Ib open-label study D5160C00006 (TATTON).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall provide AstraZeneca with an opportunity to review/comment on drafts of any publication, review article or presentation (Publication) and shall afford AstraZeneca the opportunity to review the final draft of the Publication before its submission. The PI shall give AstraZeneca up to 45 days to respond with any proposed corrections and shall delete any confidential information before submission. If requested the PI shall delay submission for an additional period, not more than 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT02454933/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT02454933/SAP_001.pdf